CLINICAL TRIAL: NCT01295723
Title: Intraoperative Boost Radiotherapy With Electrons (IOERT) Followed By Hypofractionated Whole-Breast Irradiation (WBRT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Joseph Hospital of Orange (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-003 Mobetron
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Invasive Lobular and Ductal Carcinoma
Keywords: Breast cancer; Radiation therapy; Mobetron; IOERT; IORT; Hypofractionated radiation therapy; Partial breast radiation
MeSH Terms: conditions — Carcinoma, Ductal; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraoperative Electron Radiation Therapy (Experimental): A single dose of electron irradiation given at the surgical site during the operation to remove the cancerous tumor will replace the usual 5-8 days of localized radiation. Hypofractionated Whole Breast Radiation Therapy must start within 14-56 days post operatively.
  Interventions: Radiation: Hypofractionated Whole Breast Radiation Therapy; Radiation: Intraoperative Electron Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Whole Breast Radiation Therapy — Hypofractionated Whole Breast Radiation Therapy must start within 14-56 days postoperatively (week 2-8 post-op)
  * Single reference dose per fraction: 2.7 Gy (ICRU)
  * Number of fractions: 15
  * Number of fractions per week: 5
  * Regular Radiation Therapy breaks: Weekend/ Holidays (not exceeding 7 days break)
  * Total dose: 50.5 Gy (40.5 WBRT + 10 Gy boost) Radiation: Intraoperative Electron Radiation Therapy
Radiation: Intraoperative Electron Radiation Therapy — Intraoperative Electron Radiation Therapy (IOERT) is delivered after completion of the lumpectomy and sentinel node procedure. IOERT is performed on mobile or fixed linac with variable electron energies in the range of 4-12 MeV
  Other Names: Mobetron

SUMMARY:
Hypofractionated intraoperative boost (HIOB) is defined as hypofractionated WBRT (40.5 Gy in 2.7 Gy per fraction) preceded by an intraoperative boost to the tumor bed (10 Gy IOERT). The HIOB study concept will test whether such a combined schedule is superior or iso-effective standard RT in terms of local control and cosmetic outcome.

DETAILED DESCRIPTION:
The purpose of this research study is to find out the effects (good and bad) of adding a dose of radiation to the area of the cancer during surgery to whole breast radiation therapy (WBRT) after surgery. IOERT is the application of electron radiation directly to the residual tumor or tumor bed during cancer surgery. WBRT is a type of radiation therapy used to treat patients who have cancer in the breast covering the entire breast tissue. Both immediate and long-term effects will be measured.

For patients with certain types of breast cancer, one standard treatment is removal of the area of cancer and a small amount of normal tissue around it followed by breast radiation. The radiation treatment in this situation usually lasts 3 to 5 1/2 weeks of WBRT followed by 5-8 daily radiation treatments at the site where the lump was removed called a "boost". During this study, the single dose of electron irradiation (IOERT) given at the surgical site during the operation will replace the usual 5-8 days of localized radiation and the whole breast radiation will last 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven invasive breast carcinoma (ductal and lobular)
* Age > 40 years
* Karnofsky performance status >70%
* Single discrete tumor or focal microcalcifications that can be imaged on a specimen radiograph or multifocal disease within the same quadrant with a maximum dimension of 4 cm (invasive foci)
* Nodal Status: NO-1
* Clear surgical margins: R0; min 2mm. Re-excision after IOERT is permitted but not required to achieve (-) margin.
* All grades G1 - G3
* Any hormonal receptor and Her-2 status
* Informed consent

Exclusion Criteria:

* In-situ Carcinoma without invasive component or multifocal disease > 4 cm
* Tumor stage: T3 or 4
* Nodal Status > N1 pathologically
* Surgical margins < 2mm
* Multicentricity
* Previous radiotherapy to the involved breast
* Karnofsky Index < 70%
* Mixed connective tissue diseases e.g. rheumatoid polyarthritis, thromboangitis obliterans, systemic lupus.
* Distant metastases
* Unable to provide written consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of acute and late toxicity | 5 years
  Assessment of acute toxicity of breast irradiation according to CTC-toxicity Scoring - systems:
  * At the end of Radiation Therapy
  * At time of first follow-up investigation (week 8 - 10)
  Assessment of late toxicity according to NSABP scoring - systems at 6, 12, 24, 36, 48, and 60 months

SECONDARY OUTCOMES:
Cosmetic Evaluation | 5 years
  Assessment of cosmetic outcome according to 5-point scoring system
  * Before Whole Breast Radiation Therapy
  * Not earlier than 7 months after Whole Breast Radiation Therapy
  * At yearly follow-up (photodocumentation in standardized positions) for 5 years.
Disease Free Survival | 5 years
  Recurrence assessments as documented at post-op follow-ups per protcol.
Overall Survival | 5 Years
  The length of time from the start of treatment to death within the 5 year period.

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Forouzannia, M.D., Principal Investigator — The Center for Cancer Prevention & Treatment at St. Joseph Hospital of Orange
Locations (1):
- St. Joseph Hospital of Orange, Orange, California, United States